CLINICAL TRIAL: NCT00696800
Title: A Phase III, Randomized, Double-Blind, Active-Controlled, Non-Inferiority Clinical Trial to Investigate the Efficacy and Safety of a Single Injection of Org 36286 (Corifollitropin Alfa) to Induce Multifollicular Development for Controlled Ovarian Stimulation Using Daily Recombinant FSH as Reference
Brief Title: A Study to Investigate the Efficacy and Safety of a Single Injection of Corifollitropin Alfa (Organon 36286) for Ovarian Stimulation Using Daily Recombinant Follicle Stimulating Hormone (FSH) as Reference (P05787)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05787; 2004-004771-11 (EudraCT Number); 38819 (Other: Organon); 8962-011 (Other: Merck)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2022-02

CONDITIONS: In Vitro Fertilization
Keywords: Infertility; Pharmacological effect of drugs; Hormones; Hormone substitutes and hormone antagonists; Pharmacological actions; Randomized; Multi-center; Multi-national; Double-blind; Active-controlled; Non-inferiority
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta; Glycoprotein Hormones, alpha Subunit; ganirelix; Chorionic Gonadotropin; Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 150 µg Corifollitropin Alfa (Experimental): Participants received a single subcutaneous (SC) injection of 150 µg Corifollitropin Alfa (org 36286) on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections from Stimulation Days 1 to 7 with placebo-recFSH; followed by daily SC injections with 200 IU recFSH up to the day of hCG. Daily SC injections of Ganirelix were administered from Stimulation Day 5 to the day of hCG; at which time a single dose of hCG was given when 3 follicles >= 17 mm. On the day of oocyte pick up (OPU) daily doses of progesterone were started and continued for up to 6 weeks or menses.
  Interventions: Drug: Corifollitropin alfa; Drug: Placebo RecFSH / follitropin beta; Biological: RecFSH / Follitropin beta (Days 8 to hCG); Drug: Ganirelix; Biological: hCG; Biological: Progesterone
- 200 IU recFSH (Active Comparator): Participants received a single SC injection of placebo Corifollitropin Alfa on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections with 200 IU recFSH from Stimulation Days 1 to 7; followed by daily SC injections with 200 IU recFSH up to the day of hCG. Daily SC injections of Ganirelix were given from Stimulation Day 5 to the day of hCG; at which time a single dose of hCG was administered when 3 follicles >= 17 mm. On the day of OPU daily doses of progesterone were started and continued for up to 6 weeks or menses.
  Interventions: Biological: RecFSH / Follitropin beta (Days 1 to 7); Drug: Placebo Corifollitropin alfa; Biological: RecFSH / Follitropin beta (Days 8 to hCG); Drug: Ganirelix; Biological: hCG; Biological: Progesterone

INTERVENTIONS:
Drug: Corifollitropin alfa — On the morning of day 2 or 3 of the menstrual cycle (Stimulation Day 1), a single SC injection of 150 μg (0.5 mL) Corifollitropin Alfa was administered in the abdominal wall.
  Other Names: MK-8962; SCH 900962; Org 36286
  Arms: 150 µg Corifollitropin Alfa
Biological: RecFSH / Follitropin beta (Days 1 to 7) — Daily SC injections with 200 IU fixed dose recFSH were started on Stimulation Day 1 and continued up to and including Stimulation Day 7.
  Other Names: Puregon / Follistim AQ Cartridge
  Arms: 200 IU recFSH
Drug: Placebo Corifollitropin alfa — Pre-filled syringe containing an identical solution when compared to Corifollitropin Alfa. On the morning of day 2 or 3 of the menstrual cycle (Stimulation Day 1), a single SC injection was administered in the abdominal wall.
  Arms: 200 IU recFSH
Drug: Placebo RecFSH / follitropin beta — Identical ready-for-use solution, but without the active ingedient, supplied in cartridges for SC injection with the Follistim Pen. Daily SC injections were started on Stimulation Day 1 and continued up to and including Stimulation Day 7.
  Arms: 150 µg Corifollitropin Alfa
Biological: RecFSH / Follitropin beta (Days 8 to hCG) — From Stimulation Day 8 onwards a daily SC dose of 200 IU recFSH was administered up to and including the Day of hCG.
  Other Names: Puregon / Follistim AQ Cartridge
Drug: Ganirelix — On Stimulation Day 5 a daily SC injection of 0.25 mg was started, which continued up to and including the day of hCG
  Other Names: Orgalutran/ Ganirelix Acetate Injection
Biological: hCG — When 3 follicles >= 17 mm were observed by USS, a single dose of 10,000 IU/USP hCG was administered; or, for those at risk for Ovarian Hyperstimulation Syndrome (OHSS), a lower dose of 5,000 IU/USP
  Other Names: Pregnyl / urinary hCG
Biological: Progesterone — On the day of OPU, luteal phase support was started by administering micronized progesterone of at least 600 mg/day vaginally, or at least 50 mg/day intramuscular (IM), which continued for at least 6 weeks, or up to menses.

SUMMARY:
To investigate the efficacy and safety of a single injection of 150 μg Corifollitropin Alfa (Organon 36286) to induce multifollicular development for controlled ovarian stimulation using daily recombinant FSH (recFSH) as a reference. The primary hypothesis is that a single injection of Corifollitropin Alfa is non-inferior to daily treatment with recFSH in initiating multifollicular growth.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-controlled, non-inferiority clinical trial investigating the efficacy and safety of a new treatment regimen with Corifollitropin Alfa, a recombinant gonadotropin applied to initiate and sustain follicular stimulation in controlled ovarian stimulation for Assisted Reproductive Technology (ART). For this regimen, participants receive a single injection of Corifollitropin Alfa and one week later, treatment is continued with daily recFSH up to the day of triggering final oocyte maturation. In the reference group participants receive daily injections of recFSH up to the day of triggering final oocyte maturation. Non-inferiority in ongoing pregnancy rates (assessed at least 10 weeks after embryo transfer) will be the primary endpoint for this trial. The number of oocytes retrieved will be analyzed as co-primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Females of couples with an indication for Controlled Ovarian Stimulation (COS) and in-vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI);
* >=18 and <=36 years of age at the time of signing informed consent;
* Body weight > 60 and <=90 kg and body mass index (BMI) >=18 and <=32 kg/m^2;
* Normal menstrual cycle length: 24-35 days;
* Availability of ejaculatory sperm (use of donated and/or cryopreserved sperm is allowed);
* Willing and able to sign informed consent.

Exclusion Criteria:

* History of/or any current (treated) endocrine abnormality;
* History of ovarian hyper-response or ovarian hyperstimulation syndrome

(OHSS);

* History of/or current polycystic ovary syndrome (PCOS);
* More than 20 basal antral follicles <11 mm (both ovaries combined) as measured on ultrasound scan (USS) in the early follicular phase (menstrual cycle day 2-5);
* Less than 2 ovaries or any other ovarian abnormality (including endometrioma > 10 mm; visible on USS);
* Presence of unilateral or bilateral hydrosalphinx (visible on USS);
* Presence of any clinically relevant pathology affecting the uterine cavity or fibroids >=5 cm;
* More than three unsuccessful IVF cycles since the last established ongoing pregnancy (if applicable);
* History of non- or low ovarian response to FSH/ human menopausal gonadotropin (hMG) treatment;
* History of recurrent miscarriage (3 or more, even when unexplained);
* FSH > 12 IU/L or LH > 12 IU/L as measured by the local laboratory (sample taken during the early follicular phase: menstrual cycle day 2-5);
* Any clinically relevant abnormal laboratory value based on a sample taken during the screening phase;
* Contraindications for the use of gonadotropins (e.g. tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, ovarian cysts);
* Recent history of/or current epilepsy, human immunodeficiency virus (HIV) infection, diabetes, cardiovascular, gastro-intestinal, hepatic, renal or pulmonary disease;
* Abnormal karyotyping of the patient or her partner (if karyotyping is performed);
* Smoking more than 5 cigarettes per day;
* History or presence of alcohol or drug abuse within 12 months prior to signing informed consent;
* Previous use of Org 36286;
* Use of hormonal preparations within 1 month prior to randomization;
* Hypersensitivity to any of the concomitant medication prescribed as part of the treatment regimen in this protocol;
* Administration of investigational drugs within three months prior to signing informed consent.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1509 (Actual)
Dates: Start 2006-06-27 (Actual); Primary Completion 2007-11-19 (Actual); Study Completion 2008-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lawrenz B, Beligotti F, Engelmann N, Gates D, Fatemi HM. Impact of gonadotropin type on progesterone elevation during ovarian stimulation in GnRH antagonist cycles. Hum Reprod. 2016 Nov;31(11):2554-2560. doi: 10.1093/humrep/dew213. Epub 2016 Sep 12. PMID 27619773
- [Derived] Zandvliet AS, Prohn M, de Greef R, van Aarle F, McCrary Sisk C, Stegmann BJ. Impact of patient characteristics on the pharmacokinetics of corifollitropin alfa during controlled ovarian stimulation. Br J Clin Pharmacol. 2016 Jul;82(1):74-82. doi: 10.1111/bcp.12939. Epub 2016 May 31. PMID 26991902
- [Derived] Griesinger G, Verweij PJ, Gates D, Devroey P, Gordon K, Stegmann BJ, Tarlatzis BC. Prediction of Ovarian Hyperstimulation Syndrome in Patients Treated with Corifollitropin alfa or rFSH in a GnRH Antagonist Protocol. PLoS One. 2016 Mar 7;11(3):e0149615. doi: 10.1371/journal.pone.0149615. eCollection 2016. PMID 26950065
- [Derived] Broekmans FJ, Verweij PJ, Eijkemans MJ, Mannaerts BM, Witjes H. Prognostic models for high and low ovarian responses in controlled ovarian stimulation using a GnRH antagonist protocol. Hum Reprod. 2014 Aug;29(8):1688-97. doi: 10.1093/humrep/deu090. Epub 2014 Jun 5. PMID 24903202
- [Derived] Leader A, Devroey P, Witjes H, Gordon K. Corifollitropin alfa or rFSH treatment flexibility options for controlled ovarian stimulation: a post hoc analysis of the Engage trial. Reprod Biol Endocrinol. 2013 Jun 11;11:52. doi: 10.1186/1477-7827-11-52. PMID 23758821
- [Derived] Fauser BC, Alper MM, Ledger W, Schoolcraft WB, Zandvliet A, Mannaerts BM; Engage Investigators. Pharmacokinetics and follicular dynamics of corifollitropin alfa versus recombinant FSH during ovarian stimulation for IVF. Reprod Biomed Online. 2010 Nov;21(5):593-601. doi: 10.1016/j.rbmo.2010.06.032. Epub 2010 Jun 30. PMID 20843746
- [Derived] Devroey P, Boostanfar R, Koper NP, Mannaerts BM, Ijzerman-Boon PC, Fauser BC; ENGAGE Investigators. A double-blind, non-inferiority RCT comparing corifollitropin alfa and recombinant FSH during the first seven days of ovarian stimulation using a GnRH antagonist protocol. Hum Reprod. 2009 Dec;24(12):3063-72. doi: 10.1093/humrep/dep291. Epub 2009 Aug 14. PMID 19684043

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1509 randomized participants, 1506 received treatment with either Corifollitropin Alfa or recFSH (Intent-to Treat population [ITT]).
Groups:
- 150 µg Corifollitropin Alfa: Participants received a single subcutaneous (SC) injection of 150 µg Corifollitropin Alfa on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections from Stimulation Days 1 to 7 with placebo-recombinant Follicle Stimulating Hormone (recFSH); followed by daily SC injections with 200 IU recFSH up to the day of human Chorionogonadotropin (hCG); multiple daily SC injections of Ganirelix were given from Stimulation Day 5 to the day of hCG; a single dose of hCG was administered when 3 follicles >= 17 mm were observed; and on the day of oocyte pick up (OPU) daily doses of progesterone were started and continued for up to 6 weeks or menses.
- 200 IU recFSH: Participants received a single SC injection of placebo Corifollitropin Alfa on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections with 200 IU recFSH from Stimulation Days 1 to 7; followed by daily SC injections with 200 IU recFSH up to the day of hCG; multiple daily SC injections of Ganirelix were given from Stimulation Day 5 to the day of hCG; single dose of hCG was administered when 3 follicles >= 17 mm were observed; and on the day of OPU daily doses of progesterone were started and continued for up to 6 weeks or menses.
Period: Overall Study
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Started | 757 | 752
Treated (ITT) | 756 (The ITT group) | 750 (The ITT group)
Completed | 672 (Participants who had embryos transferred) | 704 (Participants who had embryos transferred)
Not Completed | 85 | 48
Not completed — Adverse Event | 16 | 3
Not completed — Insufficient compliance with medication | 2 | 1
Not completed — Insufficient ovarian response on Day 8 | 4 | 1
Not completed — Insufficient ovarian response | 4 | 1
Not completed — Risk Ovarian Hyperstimulation Syndrome | 8 | 2
Not completed — Too high ovarian response | 6 | 1
Not completed — No/too few/bad quality oocytes | 4 | 3
Not completed — No/abnormal fertilization | 11 | 13
Not completed — No/too few/bad quality embryos | 24 | 18
Not completed — Other Reasons | 5 | 3
Not completed — Not treated | 1 | 2

BASELINE CHARACTERISTICS:
Population: The ITT group consisting of randomized participants treated with Corifollitropin Alfa or recFSH
Groups:
- 150 µg Corifollitropin Alfa: Participants received a single SC injection of 150 µg Corifollitropin Alfa on day 2 or 3 of the menstrual cycle (Stimulation Day 1); 7 daily SC injections from Stimulation Days 1 to 7 with placebo-recFSH; followed by daily SC injections with 200 IU recFSH up to the day of hCG; multiple daily SC injections of Ganirelix were given from Stimulation Day 5 to the day of hCG; a single dose of hCG was administered when 3 follicles >= 17 mm were observed; and on the day of OPU daily doses of progesterone were started and continued for up to 6 weeks or menses.
- Total: Total of all reporting groups
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH | Total
Number analyzed (Participants) | 756 | 750 | 1506
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.5 (3.3) | 31.5 (3.2) | 31.5 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 756 | 750 | 1506
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Ongoing Pregnancy (Ongoing Pregnancy Rate)
Description: An ongoing pregnancy is a fetus with heart activity at least 10 weeks after embryo transfer as assessed by Ultrasound Scan (USS) or Doppler or is confirmed by live birth. The ongoing pregnancy rate is 100 times the number of participants with an ongoing pregnancy after embryo transfer, divided by the total number of participants who started treatment. Calculations were made per attempt, meaning that participants who did not have embryo transfers were considered not pregnant.
Time Frame: Assessed at least 10 weeks after embryo transfer (up to 1 year)
Population: Intent to Treat (ITT) population consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 756 | 750
Percentage of participants | 39.0 | 38.1
Statistical Analysis 1: Comparison: 150 µg Corifollitropin Alfa vs 200 IU recFSH; Test type: Non-Inferiority or Equivalence — Treatment groups were formally compared with a generalized linear model for the ongoing pregnancy rate which included factors for treatment group, age at randomization, and region. A pre-defined non-inferiority margin of 8% was applied; Risk Difference (RD) = 1.1, 95% CI 2-sided [-3.8 to 5.9]

2. Primary Outcome: Mean Number of Oocytes Retrieved
Description: Up to 36 hours after receiving hCG, cumulus-oocyte-complexes were retrieved. Mean numbers retrieved were calculated per attempt, meaning that if a participant did not reach this stage in In Vitro Fertilization (IVF) treatment, zero values were imputed.
Time Frame: Up to 36 hours after administration of hCG (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to.
Measure: Mean (Standard Deviation); unit: Number of oocytes
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 756 | 750
Number of oocytes | 13.8 (8.3) | 12.6 (6.8)
Statistical Analysis 1: Comparison: 150 µg Corifollitropin Alfa vs 200 IU recFSH; Test type: Non-Inferiority or Equivalence — Equivalence margins of -3 and +5 were applied for the difference in number of oocytes. If the 95% confidence interval of the difference exceeded -3 or +5 oocytes, then Corifollitropin Alfa treatment was not considered equivalent to the reference treatment (recFSH); p = 0.001, ANOVA — Treatment groups were formally compared including covariates treatment group, age and center; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.5 to 1.9]

3. Secondary Outcome: Median Amount of Recombinant FSH Needed to Induce Multifollicular Development Starting at Day 1
Description: The amount of recFSH administered for a participant to reach 3 follicles >= 17 mm, starting from treatment Day 1 onwards.
Time Frame: From Day 1 to day of hCG treatment (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants with hCG injection.
Measure: Median (Full Range); unit: IU
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 733 | 741
IU | 400 [0 to 2000] | 1800 [400 to 2800]

4. Secondary Outcome: Median Amount of Recombinant FSH Needed to Induce Multifollicular Development Starting at Day 8
Description: The amount of recFSH administered for a participant to reach 3 follicles >= 17 mm, starting from treatment Day 8 onwards.
Time Frame: From Day 8 to Day of hCG treatment (up to 1 year)
Population: as for outcome 3
Measure: Median (Full Range); unit: IU
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 733 | 741
IU | 400 [0 to 2000] | 400 [0 to 1400]

5. Secondary Outcome: Serum FSH Levels During Stimulation
Description: Mean serum FSH are presented over one Controlled Ovarian Stimulation (COS) cycle: from Day 1 (Pre-dose) up to the day of hCG treatment.
Time Frame: Up to day of hCG treatment (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa (Cori Alfa) or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants who had FSH data available.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 732 | 724
IU/L
  Day 1 (Pre-dose) (Cori. Alfa N=732; recFSH N=724) | 6.70 (2.05) | 6.60 (1.86)
  Day 5 (Cori. Alfa N=725; recFSH N=722) | 23.49 (6.22) | 11.61 (3.40)
  Day 8 (Cori. Alfa N=708; recFSH N=678) | 11.76 (3.18) | 11.59 (2.65)
  Day of hCG (Cori. Alfa N=698; recFSH N=708) | 12.54 (3.35) | 11.59 (2.80)

6. Secondary Outcome: Serum Luteinizing Hormone (LH) Levels During Stimulation
Description: Mean serum LH levels are presented over one COS cycle: from Day 1 (Pre-dose) up to the day of hCG treatment.
Time Frame: Up to day of hCG treatment (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa (Cori Alfa) or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants who had LH data available.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 732 | 724
IU/L
  Day 1 (Pre-dose) (Cori. Alfa N=732; recFSH N=724) | 4.80 (2.02) | 4.67 (1.82)
  Day 5 (Cori. Alfa N=725; recFSH N=722) | 3.62 (4.60) | 2.23 (2.92)
  Day 8 (Cori. Alfa N=708; recFSH N=678) | 1.29 (1.80) | 2.05 (1.80)
  Day of hCG (Cori. Alfa N=698; recFSH N=708) | 1.38 (1.79) | 1.86 (1.63)

7. Secondary Outcome: Serum Estradiol (E2) Levels During Stimulation
Description: Mean serum E2 levels are presented over one COS cycle: from Day 1 (Pre-dose) up to the day of hCG treatment.
Time Frame: Up to day of hCG treatment (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa (Cori Alfa) or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants who had E2 data available.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 732 | 724
pmol/L
  Day 1 (Pre-dose) (Cori. Alfa N=732; recFSH N=724) | 126.13 (39.17) | 124.79 (37.11)
  Day 5 (Cori. Alfa N=725; recFSH N=722) | 1859.39 (1224.78) | 1392.97 (895.66)
  Day 8 (Cori. Alfa N=708; recFSH N=678) | 3700.92 (2837.41) | 3750.96 (2600.03)
  Day of hCG (Cori. Alfa N=698; recFSH N=708) | 5486.67 (3461.92) | 5154.88 (2999.48)

8. Secondary Outcome: Serum Progesterone (P) Levels During Stimulation
Description: Mean serum P levels are presented over one COS cycle: from Day 1 (Pre-dose) up to day of hCG treatment
Time Frame: Up to day of hCG treatment (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa (Cori Alfa) or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants who had P data available.
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 732 | 724
nmol/mL
  Day 1 (Pre-dose) (Cori. Alfa N=732; recFSH N=724) | 1.80 (1.28) | 1.85 (1.42)
  Day 5 (Cori. Alfa N=725; recFSH N=722) | 2.13 (1.97) | 1.61 (0.87)
  Day 8 (Cori. Alfa N=708; recFSH N=678) | 1.95 (1.06) | 2.64 (1.21)
  Day of hCG (Cori. Alfa N=698; recFSH N=708) | 3.20 (4.88) | 3.16 (1.47)

9. Secondary Outcome: Serum Inhibin-B Levels During Stimulation
Description: Mean serum Inhibin-B levels are presented over one COS cycle: from Day 1 (Pre-dose) up to day of hCG treatment
Time Frame: Up to day of hCG treatment (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa (Cori Alfa) or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants who had Inhibin-B data available.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 736 | 724
pg/mL
  Day 1 (Pre-dose) (Cori. Alfa N=736; recFSH N=724) | 52.78 (29.29) | 52.95 (27.02)
  Day 5 (Cori. Alfa N=731; recFSH N=724) | 488.54 (380.13) | 493.86 (329.71)
  Day 8 (Cori. Alfa N=713; recFSH N=679) | 578.21 (508.40) | 642.27 (464.05)
  Day of hCG (Cori. Alfa N=704; recFSH N=710) | 608.35 (489.52) | 612.19 (435.26)

10. Secondary Outcome: Number of Follicles Categorized by Size on Stimulation Day 1
Description: Ovaries were assessed during stimulation by ultrasonographic investigation (USS), and the mean number of follicles are categorized by their size.
Time Frame: On Day 1 of treatment (up to 1 year)
Population: ITT population (consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to) with USS data available on Stimulation Day 1.
Measure: Mean (Standard Deviation); unit: Number of follicles
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 714 | 714
Number of follicles
  >=11 mm | 0.1 (0.3) | 0.1 (0.4)
  >=15 mm | 0.0 (0.2) | 0.0 (0.2)
  >=17 mm | 0.0 (0.2) | 0.0 (0.2)

11. Secondary Outcome: Number of Follicles Categorized by Size on Stimulation Day 5
Description: Ovaries were assessed during stimulation by USS, and the mean number of follicles are categorized by their size.
Time Frame: On Day 5 of treatment (up to 1 year)
Population: ITT population (consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to) with USS data available on Stimulation Day 5.
Measure: Mean (Standard Deviation); unit: Number of follicles
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 748 | 749
Number of follicles
  >=11 mm | 4.4 (3.8) | 4.7 (3.9)
  >=15 mm | 0.3 (0.7) | 0.4 (0.9)
  >=17 mm | 0.1 (0.3) | 0.1 (0.4)

12. Secondary Outcome: Number of Follicles Categorized by Size on Stimulation Day 8
Description: Ovaries were assessed during stimulation by USS, and the mean number of follicles are categorized by their size.
Time Frame: On Day 8 of treatment (up to 1 year)
Population: ITT population (consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to) with USS data available on Stimulation Day 8.
Measure: Mean (Standard Deviation); unit: Number of follicles
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 729 | 703
Number of follicles
  >=11 mm | 12.8 (6.7) | 11.6 (6.0)
  >=15 mm | 5.0 (4.6) | 5.2 (4.1)
  >=17 mm | 2.1 (2.9) | 2.5 (2.8)

13. Secondary Outcome: Number of Follicles Categorized by Size on the Day of hCG
Description: Ovaries were assessed during stimulation by USS, and the mean number of follicles are categorized by their size.
Time Frame: Day of HCG treatment (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants with hCG injection and with USS data available.
Measure: Mean (Standard Deviation); unit: Number of follicles
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 723 | 734
Number of follicles
  >=11 mm | 16.0 (7.0) | 13.9 (6.1)
  >=15 mm | 9.6 (4.8) | 8.7 (4.0)
  >=17 mm | 5.7 (3.2) | 5.6 (2.9)

14. Secondary Outcome: Number of Cumulus-oocyte-complexes
Description: Prior to IVF the mean number of cumulus-oocyte-complexes used for IVF was assessed
Time Frame: Up to 36 hours after administration of hCG (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants who underwent IVF.
Measure: Mean (Standard Deviation); unit: Number of cumulus-oocyte complexes
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 242 | 240
Number of cumulus-oocyte complexes | 13.6 (8.2) | 12.8 (7.0)

15. Secondary Outcome: Number of Oocytes Assessed Prior to Intracytoplasmic Sperm Injection (ICSI)
Description: The number of oocytes used for ICSI was assessed, and categorized based on their quality
Time Frame: Up to 36 hours after administration of hCG (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa (Cori Alfa) or recFSH, and grouped according to the treatment they were randomized to. For participants who had ICSI; but also includes 3 participants whose oocytes were assessed, but ICSI was not performed.
Measure: Mean (Standard Deviation); unit: Number of oocytes
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 413 | 417
Number of oocytes
  Total | 13.8 (7.7) | 12.2 (6.4)
  Metaphase I | 1.1 (1.5) | 0.9 (1.3)
  Metaphase II | 10.8 (6.5) | 9.2 (5.1)
  Germinal vesicles | 1.4 (1.9) | 1.7 (2.2)

16. Secondary Outcome: Percentage of Fertilized Oocytes (Fertilization Rate)
Description: The fertilization rate is 100 times the number of fertilized 2 pro-nuclei (2PN) oocytes obtained, divided by the number of oocytes fertilized by IVF or ICSI
Time Frame: Up to 18 hours after start of fertilization (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to.Restricted to participants with IVF and/or ICSI.
Measure: Mean (Standard Deviation); unit: Percentage of fertilized oocytes
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 728 | 737
Percentage of fertilized oocytes | 66.0 (23.5) | 67.6 (22.9)

17. Secondary Outcome: Number of Embryos Obtained on Day 3 Categorized by Quality
Description: Embryos obtained on Day 3 were categorized by their qualiity as follows: Grade 1: excellent: No fragmentation, 6-10 cells, and equal blastomere size taking the impact of cell division into account. Grade 2: good: < 20% fragmentation, 6-10 cells, and equal blastomere size taking the impact of cell division into account. Grade 3: fair: 20-50% fragmentation and/or less than 6 cells and/or multinucleation (if observed). Other Grade: Embryos that do not qualify as Grades 1, 2 or 3. Grades 1 and 2 are considered good quality.
Time Frame: Post fertilization Day 3 (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants with IVF and/or ICSI, and excludes those who had embryos transferred or cryopreserved before Day 3.
Measure: Mean (Standard Deviation); unit: Number of embryos
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 714 | 729
Number of embryos
  Total | 8.4 (5.5) | 7.5 (4.8)
  Good Quality | 4.7 (4.3) | 4.5 (3.9)
  Grade 1 | 2.6 (3.4) | 2.5 (3.4)
  Grade 2 | 2.1 (2.5) | 2.0 (2.3)
  Grade 3 | 2.4 (2.6) | 2.0 (2.3)
  Other Grade | 1.4 (2.2) | 1.1 (2.1)

18. Secondary Outcome: Number of Embryos Transferred on Day 3
Description: After fertilization, the mean number of embryos transferred on Day 3 were assessed. Total and good quality embryos are presented, with good quality embryos, Grades 1 and 2, defined as the following: Grade 1: excellent: No fragmentation, 6-10 cells, and equal blastomere size taking the impact of cell division into account. Grade 2: good: < 20% fragmentation, 6-10 cells, and equal blastomere size taking the impact of cell division into account.
Time Frame: Post fertilization Day 3 (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants with embryo transfer.
Measure: Mean (Standard Deviation); unit: Number of embryos
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 672 | 704
Number of embryos
  Total | 1.7 (0.4) | 1.7 (0.4)
  Good Quality | 1.4 (0.7) | 1.4 (0.7)

19. Secondary Outcome: Percentage of Gestational Sacs (Implantation Rate)
Description: The implantation rate is 100 times the number of gestational sacs assessed by USS after embryo transfer, divided by the number of embryos transferred.
Time Frame: Up to 6 weeks after embryo transfer (up to 1 year)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percentage of gestational sacs
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 672 | 704
Percentage of gestational sacs | 36.2 (41.6) | 32.2 (40.1)

20. Secondary Outcome: Percentage of Participants With a Miscarriage (Miscarriage Rate) Per Clinical Pregnancy
Description: The miscarriage rate is 100 times the number of miscarriages, divided by the number of clinical pregnancies assessed by USS. A clinical pregnancy is the presence of at least one gestational sac or confirmed by live birth.
Time Frame: Up to day of miscarriage (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants with a clinical pregnancy.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 322 | 308
Percentage of participants | 8.4 | 6.8

21. Secondary Outcome: Percentage of Participants With a Miscarriage (Miscarriage Rate) Per Vital Pregnancy
Description: The miscarriage rate is 100 times the number of miscarriages, divided by the number of vital pregnancies assessed by USS. A vital pregnancy is the presence of at least one fetus with heart activity.
Time Frame: Up to day of miscarriage (up to 1 year)
Population: ITT population consisting of all randomized participants who were treated with Corifollitropin Alfa or recFSH, and grouped according to the treatment they were randomized to. Restricted to participants with a vital pregnancy.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 302 | 293
Percentage of participants | 2.3 | 2.0

22. Secondary Outcome: Percentage of Participants With a Biochemical Pregnancy (Pregnancy Rate) Per Attempt
Description: Biochemical pregnancy was assessed by measuring serum or urinary hCG. Per attempt means that if a participant did not reach the stage of pregnancy assessment zero values were imputed. The pregnancy rate is 100 times the number of participants with pregnancies detected, divided by the number of participants assessed.
Time Frame: Two weeks after embryo transfer (up to 1 year)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 756 | 750
Percentage of participants | 48.1 | 46.9

23. Secondary Outcome: Percentage of Participants With a Biochemical Pregnancy (Pregnancy Rate) Per Embryo Transfer
Description: Biochemical pregnancy was assessed for participants who had embryo transfer by measuring serum or urinary hCG. The pregnancy rate is 100 times the number of participants with pregnancies detected, divided by the number of participants assessed.
Time Frame: Two weeks after embryo transfer (up to 1 year)
Population: as for outcome 18
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Number analyzed (Participants) | 672 | 704
Percentage of participants | 54.2 | 50.0

ADVERSE EVENTS:
Time Frame: Up to 10 weeks after embryo transfer (up to 1 year)
Description: The All-Subjects-Treated (AST) group. AST is based on the treatment actually received. Two participants randomized to the 150 µg Corifollitropin Alfa treatment group were actually treated with 200 IU recFSH, whereas one participant randomized to the 200 IU recFSH treatment group was actually treated with 150 µg Corifollitropin Alfa.
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU recFSH
Serious Adverse Events (participants affected / at risk) | 35/755 | 30/751
Other Adverse Events (participants affected / at risk) | 403/755 | 383/751
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 µg Corifollitropin Alfa (N=755) | 200 IU recFSH (N=751)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 6 (6)
Heterotopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3)
Haematosalpinx (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 14 (14) | 9 (9)
Ovarian torsion (Reproductive system and breast disorders) | 2 (2) | 4 (4)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
Selective abortion (Surgical and medical procedures) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 µg Corifollitropin Alfa (N=755) | 200 IU recFSH (N=751)
Nausea (Gastrointestinal disorders) | 77 (81) | 82 (100)
Fatigue (General disorders) | 43 (47) | 37 (41)
Post procedural complication (Injury, poisoning and procedural complications) | 53 (65) | 52 (59)
Post procedural discomfort (Injury, poisoning and procedural complications) | 43 (47) | 43 (46)
Procedural pain (Injury, poisoning and procedural complications) | 173 (182) | 157 (169)
Headache (Nervous system disorders) | 81 (107) | 116 (153)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 75 (104) | 61 (83)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 53 (69) | 47 (55)
Pelvic discomfort (Reproductive system and breast disorders) | 89 (128) | 87 (106)
Pelvic pain (Reproductive system and breast disorders) | 91 (127) | 92 (115)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be based on data validated and released by the Sponsor. Any scientific paper, presentation or other communication concerning this clinical trial will first be submitted to the Sponsor at least six weeks before publication or presentation. The Sponsor shall have the right to make its consent conditional upon proper representation of the interpretation of both the Sponsor and the investigator(s) in the discussion of the data in such communications.